CLINICAL TRIAL: NCT05509894
Title: Post Marketing Surveillance (PMS) Study for Ngenla Prefilled Pen in Pediatric Patients Who Have Endogenous Growth Failure Due to an Inadequate Secretion of Endogenous Growth Hormone in Korea
Brief Title: Korean Post-marketing Surveillance Ngenla® Pre-filled Pen Injection for the Treatment of Pediatric Patients With Growth Disturbance Due to Insufficient Secretion of Growth Hormone
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0311016
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: Pediatric Growth Hormone Deficiency; Somatrogon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving Ngenla: Participants receiving Ngenla according to label
  Interventions: Drug: Ngenla

INTERVENTIONS:
Drug: Ngenla — As provided in real world practice

SUMMARY:
This non-interventional study will be performed by design of post-marketing surveillance (PMS) as an additional pharmacovigilance activity of the Risk Management Plan (RMP) for Ngenla® pre-filled pen injection, which is required by the Ministry of Food and Drug Safety (MFDS) according to the local regulation. This post-marketing surveillance will investigate the safety and effectiveness of Ngenla® pre-filled pen injection as the treatment of children and adolescents from 3 years of age with growth disturbance due to insufficient secretion of growth hormone during 6 years under the setting of routine practice in Korea.

ELIGIBILITY:
Inclusion Criteria:

- 1. Children and adolescents from 3 years of age with growth disturbance due to insufficient secretion of growth hormone who have received treatment with somotarogon or have been determined to start treatment with somatrogon according to the approved indications of the medicinal product;

2. Evidence of a personally signed and dated informed consent document indicating that the patient or their parent(s)/legal guardian, if applicable, have been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Patients concurrently participating in other studies involving therapeutic interventions and/or investigational products;
2. Patients who have contraindications to somatrogon as specified in the approved LPD.
3. Patients with hypersensitivity or case history to somatrogon or to any of the excipients in the product

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be performed in patients who have received at least 1 dose of Ngenla® pre-filled pen injection for the following indications as per local product label. (Treatment of children and adolescents from 3 years of age with growth disturbance due to insufficient secretion of growth hormone)
Sampling Method: Non-Probability Sample
Enrollment: 565 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | up to 28 days after last dose

SECONDARY OUTCOMES:
Change from baseline in Annualized Height Velocity in cm/year | baseline, up to 12 months
Change from baseline in Height Standard Deviation Score | baseline, up to 12 months
Change from baseline in Bone Maturation (BM) | baseline, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0311016